CLINICAL TRIAL: NCT02759263
Title: Pilot Study of Executive Function Intervention to Improve Neurodevelopmental Outcomes in Adolescents With CHD
Brief Title: Improving Neurodevelopment in Adolescents With Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Thrasher Research Fund (Other); The Children's Heart Foundation (Other)
Responsible Party: Principal Investigator, Jane W. Newburger, MD, Commonwealth Professor of Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-P00022266
Record Dates: First submitted 2016-04-22; First posted 2016-05-03 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Congenital Heart Disease; Neurodevelopment; Executive Function; Working Memory Training; Infant Open-heart Surgery
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Working Memory Intervention (Experimental): The group randomized to the Working Memory intervention will receive Cogmed computerized training of executive function and attention skills. The standard Cogmed RM will be used for this trial arm. This is a child-friendly web-based software program. The investigators will use a version of the program that contains 12 different neurocognitive tasks. Tasks become more difficult as a function of performance on a session-by-session basis. Each training session lasts 35-40 minutes, with one session to be completed per day 5 days each week for 5 weeks, for a total of 25 sessions. The program yields individual session-by-session and task-by- task training results, including the adolescents' responses, time spent on each task, and evolution curves.
  Interventions: Behavioral: Cogmed Working Memory Training
- Control group - Standard of Care (No Intervention): Adolescents randomly assigned to the control group will receive the standard of care recommended for patients with critical CHD. This includes cardiac surveillance and neurodevelopmental counseling and screening at our Cardiac Neurodevelopmental Program if needed. Once enrolled in our study, an adolescent in the control group will not receive Cogmed intervention or any other cognitive intervention that targets executive functions or ADHD symptoms until after the 3-month follow-up neurodevelopmental evaluation is performed, i.e., 5-6 months after initial enrollment. Like adolescents assigned to the intervention group, controls can continue on treatments that are already in place for other neurodevelopmental disabilities (e.g., speech therapy, occupational services).

INTERVENTIONS:
Behavioral: Cogmed Working Memory Training — Cogmed Working Memory Program will be used as a computerized home-based intervention. Families will receive a link for downloading a web-based software program. The program will be installed on a computer at a family's home by a research assistant. Parents and adolescents will be actively involved, and during the installation session, adolescents will complete several practice trials. The 25 sessions will be completed individually by the adolescent with parental supervision. For the first 5 sessions, the participant trains on the same set of games; on the 6th session and every 5th session thereafter, a new task is introduced and replaces one of the initial tasks. At the end of each session, the adolescent can play an age-appropriate computerized game as a reward. After each session, results are uploaded by parents to a secure website, to keep track of the participant's progress. Families will be contacted weekly to check program function and discuss concerns.
  Arms: Working Memory Intervention

SUMMARY:
Executive dysfunction can profoundly impact all dimensions of a child's development. Impairments in executive function are a central component of the neurodevelopmental phenotype associated with CHD, and manifest as behavioral dysregulation and problems with attention, working memory, and organization/planning abilities. Identifying effective treatment strategies is vital for providing optimal care for these patients. The Cogmed executive function intervention, an evidence-based computerized neurocognitive program, improves outcomes in several pediatric populations. The investigators propose to conduct a pilot study to evaluate its efficacy in reducing morbidities in patients with CHD. This is a single center, single blinded 2-arm randomized controlled trial to test the immediate post-treatment and 3-month follow-up efficacy of Cogmed intervention versus standard of care in adolescents with CHD.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CHD requiring open-heart surgery before age 1 year.
2. Ages 13-16 years old.
3. ≥ 6 months post-cardiac surgery.
4. Followed-up at the Cardiology clinic of Boston Children's Hospital.
5. English and/or Spanish speaking.
6. Home internet access and a computer on which the Cogmed program can be installed
7. Informed consent of parent/guardian as well as assent of child.

Exclusion Criteria:

1. Chromosomal anomalies and/or genetic syndromes.
2. Severe physical and/or sensory impairments (hearing, visual, or psychomotor).
3. IQ scores <85 at baseline
4. Confirmed diagnosis of an autism spectrum disorder or a severe developmental disorder that would prevent successful completion of the planned study testing.
5. Scheduled to undergo major cardiac interventions in the 6 months following enrollment.
6. Received, receiving, or scheduled to receive Cogmed or any other computerized behavioral training program targeting executive functions or ADHD.

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline scores at the computerized Working Memory Test from the NIH Toolbox Assessment of Neurological and Behavioral Function at post-treatment assessment (up to 2 weeks after cessation of the intervention). | Post-treatment assessment (up to 2 weeks after the cessation of the intervention)
  This standardized measure assesses the ability to process information across a series of modalities (visual-spatial and verbal), to hold this information in a short-term buffer, and to actively manipulate it mentally. It is considered an excellent composite indicator of adolescents' executive function skills, as it requires the simultaneous implementation of control of attention and working memory abilities on tasks of increasing complexity. Mean scores are automatically computed and are compared to a standardization sample of US adolescents of the same age. They are normally distributed (mean=100, SD=15).

CONTACTS AND LOCATIONS:
Overall Officials: Jane W Newburger, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Calderon J, Wypij D, Rofeberg V, Stopp C, Roseman A, Albers D, Newburger JW, Bellinger DC. Randomized Controlled Trial of Working Memory Intervention in Congenital Heart Disease. J Pediatr. 2020 Dec;227:191-198.e3. doi: 10.1016/j.jpeds.2020.08.038. Epub 2020 Aug 19. PMID 32827526